CLINICAL TRIAL: NCT06747858
Title: A Phase 2, Open-label, Multiple Ascending-Dose Study to Evaluate the Safety, Tolerability and Efficacy of ARCT-032 in People With Cystic Fibrosis
Brief Title: Safety, Tolerability and Efficacy Study of ARCT-032 in People With Cystic Fibrosis
Acronym: LunairCF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Arcturus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARCT-032-02
Record Dates: First submitted 2024-12-17; First posted 2024-12-24 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis; CFTR Gene Mutation
Keywords: CFTR; mRNA
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Multiple ascending dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Dose Level A of ARCT-032, inhaled daily for 28 days
  Interventions: Biological: ARCT-032
- Cohort 2 (Experimental): Dose Level B of ARCT-032, inhaled daily for 28 days
  Interventions: Biological: ARCT-032
- Cohort 3 (Experimental): Dose Level C of ARCT-032, inhaled daily for 28 days
  Interventions: Biological: ARCT-032

INTERVENTIONS:
Biological: ARCT-032 — CFTR mRNA formulated in lipid nanoparticles

SUMMARY:
ARCT-032-02 is a Phase 2, open-label, multicenter, multiple-ascending dose study of ARCT-032 in adults with CF who are not eligible for CFTR modulator therapy or are not taking CFTR modulators due to drug intolerance, poor response, or lack of access to modulators.

DETAILED DESCRIPTION:
This is an open-label, multiple-ascending dose study of ARCT-032 in adults with CF who are not on CFTR modulator therapy. After successful screening, eligible participants will receive nebulized ARCT-032 daily for 4 weeks, and then followed for safety for a total of 12 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Confirmed diagnosis of Cystic Fibrosis
2. Not eligible for CFTR modulator therapy, or not taking CFTR modulators for at least 60 days prior to dosing (e.g. due to intolerance, poor response, or lack of access to modulators).
3. FEV1 between 40% and 100% of predicted value

Exclusion Criteria:

1. History of illness or medical condition that might pose an additional risk or may confound study results
2. Recent moderate or severe hemoptysis
3. Recent major surgery
4. Solid organ or hematologic transplant
5. Requirement of supplemental oxygen while awake or > 2L per minute while sleeping.
6. Chronic maintenance systemic corticosteroids exceeding equivalent of daily 15 mg oral prednisone or 30 mg every other day
7. Adequate liver and kidney function as determined by lab tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity and dose relationship of adverse events | 16 weeks
  Safety and tolerability of ARCT-032 assess by determining incidence, severity and dose-relationship of AEs by dose level

SECONDARY OUTCOMES:
Pharmacokinetics | Up to 6 weeks
  Plasma concentration of ARCT-032 mRNA and lipid components
Pharmacodynamics--Lung Function | 4 weeks
  Change from baseline in FEV1
Pharmacodynamics--Cystic Fibrosis Quality of Life Questionnaire-Revised (CFQ-R) | 4 weeks
  Change from baseline in CFQ-R RSS (Respiratory Symptoms Scale) Score. Overall CFQ-R score ranges from 0-100, with higher scores indicating better health.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Arizona, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - The Cystic Fibrosis Institute, Northfield, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Vanderbilt University, Nashville, Tennessee
  - UT Health, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No